CLINICAL TRIAL: NCT01366885
Title: Study of Vitamin D to Prevent Autism in Newborn Siblings
Brief Title: Vitamin D to Prevent Autism in Newborn Siblings
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Gene Stubbs, Associate Professor Emeritus of Psychiatry and Pediatrics, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OHSU-AS-11-1-11
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Autistic Disorder
Keywords: Autism; Pregnancy; Newborn siblings
MeSH Terms: conditions — Autistic Disorder | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention during pregnancy (Experimental): 5000 IU Vitamin D3 to be given to the mother during pregnancy. 7000 IU Vitamin D3 to be given during breast feeding if breast feeding. If not breastfeeding, infant to be given 400 IU Vitamin D3 during first year of age, then increased to 1000 IU D3 until completion of research trial.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — 5000 IU D3 capsule oral/day for entire pregnancy. 7000 IU D3/day during breastfeeding. If not breast feeding, baby gets 400 IU D3/day. Baby increased to 1000 IU D3/day at one year of age.
  Other Names: Cholecalciferol

SUMMARY:
The purpose of this study is to determine whether by administering vitamin D to mothers who already have at least one child with autism and who are pregnant, that the vitamin D will prevent the recurrence of autism in the newborn sibling.

DETAILED DESCRIPTION:
The incidence of autism is increasing. Also, women of childbearing age are increasingly found to be insufficient/deficient in vitamin D. Vitamin D is a neurohormone which is important for development of the child, especially of the child's brain. The primary source of vitamin D is from the sun through one's skin. People have been avoiding the sun because of skin cancer, because of increasing Television watching, computer viewing and wearing clothes that cover most of the body. This approach will study whether making the pregnant mother, whose child is at risk for autism because of a previous child with autism, replete with vitamin D will prevent that recurrence of autism in the newborn sibling.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers who have had at least one child with autism spectrum disorder

Exclusion Criteria:

* Child with autism must not be from a syndrome such as Fragile X syndrome, Retts Syndrome
* Mother must be before the third trimester

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin G. Stubbs, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Evergreen Center, Oregon City, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Please see publication in Medical Hypotheses-88(2016) 74-78-entitled: Autism: Will vitamin D Supplementation during pregnancy and early childhood reduce the recurrence rate of autism in newborn siblings? G. Stubbs et al.

REFERENCES:
- [Background] Cannell JJ. On the aetiology of autism. Acta Paediatr. 2010 Aug;99(8):1128-30. doi: 10.1111/j.1651-2227.2010.01883.x. Epub 2010 May 19. No abstract available. PMID 20491697

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention During Pregnancy
Started | 20 (We started recruiting in February 2008 and recruited 20 mothers.)
Completed | 19 (We completed our study when the last child born had reached 36 months of age.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Mothers of at least one child with autism and pregnant before the third trimester
Arm/Group | Intervention During Pregnancy
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Females | 20
Region of Enrollment [Number; unit: participants]
  United States | 19
  Israel | 1
Mothers with at least one child with autism, and pregnant before the third trimester [Number; unit: participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Who Developed Autism
Description: The child will be screened by an Modified Checklist for Autism in Toddlers (MCHAT) interview at 18 months of age, and by a questionnaire, the Pervasive Developmental Disorder Behavioral Inventory (PDDBI) at 3 years of age to determine whether the child has developed autism or not.
Time Frame: Child assessed at 3 years of age
Population: Children who developed autism
Measure: Number; unit: Children who developed autism
Arm/Group | Intervention During Pregnancy
Number analyzed (Participants) | 19
Children who developed autism | 1

2. Secondary Outcome: Number of Mothers Who Developed Side Effects From Vitamin D
Description: Mother will be followed by blood and urine screening for hypercalcemia and hypercalciuria which is the primary side effects of too much vitamin D.
Time Frame: During pregnancy and the 3 years of the child's development
Population: The children born were assessed for whether they developed autism or not.
Measure: Number; unit: participants
Arm/Group | Intervention During Pregnancy
Number analyzed (Participants) | 19
participants | 0

ADVERSE EVENTS:
Arm/Group | Intervention During Pregnancy
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No